CLINICAL TRIAL: NCT05153980
Title: The Impact of Blood Flow Restriction Within Warm-up Routines on Performance and Muscle Stiffness.
Brief Title: The Impact of Blood Flow Restriction Within Warm-up.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: B6702021000931
Record Dates: First submitted 2021-11-15; First posted 2021-12-10 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Healthy
Keywords: Shear Wave Elastography; Blood Flow Restriction; Warm-up; Performance
MeSH Terms: interventions — Warm-Up Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blood Flow Restriction (Experimental): Incorporation of Blood Flow Restriction within the warm-up routine.
  Interventions: Device: Warm-up + Blood Flow Restriction cuff (smart-cuff pro device, acting as pressurized tourniquet)
- Control Group (Active Comparator): Warm-up routine without any special intervention (no Blood Flow Restriction).
  Interventions: Other: Warm-up

INTERVENTIONS:
Device: Warm-up + Blood Flow Restriction cuff (smart-cuff pro device, acting as pressurized tourniquet) — Blood Flow Restriction
  Other Names: Kaatsu; partial vascular occlusion
  Arms: Blood Flow Restriction
Other: Warm-up — Warm-up without any special intervention (no Blood Flow Restriction)
  Arms: Control Group

SUMMARY:
Sixty athletes will be randomized in two groups; (1) an experimental group and (2) a control group. Both groups will undergo the following procedure:

Moment 1:

1. Baseline testing: countermovement jump, 25m sprint and strength assessment of the Hamstrings and Quadriceps muscle.
2. Short warm-up (approximately 4 minutes), which will be completed with blood flow restriction cuffs (experimental group) or without (control group)
3. Post testing: same tests as performed in baseline.

Moment 2:

1. Baseline testing: stiffness measurements of the Biceps Femoris Long Head via Shear Wave Elastography.
2. Short warm-up (approximately 4 minutes), which will be completed with blood flow restriction cuffs (experimental group) or without (control group)
3. Post testing: same tests as performed in baseline.

Both moments of testing as well as the order in which the performance tests take place are randomized.

DETAILED DESCRIPTION:
Traditionally, athletes perform a warm-up program before participating in sport activities, due to its assumed beneficial effect on performance and injury prevention. However, within team sports, substitutes usually do not perform the comprehensive pre-match warm-up. In many cases, those substitute players get a very short period of time, during the game, to prepare themselves for coming on to the pitch where they immediately have to perform at a very high-intensity. Hence, this could lead to a poorer performance and a greater injury risk for those substitute players, as they did not get a decent warm-up.

Therefore, new techniques are needed in order to prepare the substitute athletes optimally in a very short period of time (often within a few minutes). Consequently, the aim of this study is to investigate whether the incorporation of Blood Flow Restriction (BFR) within a warm-up routine could be of additional value. Both performance parameters and muscle stiffness will be evaluated. As Hamstring strain Injuries (HSI) are common within sports encompassing high-speed running, this muscle group will be investigated on muscle stiffness as a representation of the interventional effect on muscle stiffness. Athletes will be randomized in two groups of 30 participants (anticipated); (1) an experimental group and (2) a control group. Both groups will perform baseline testing (5x Countermovement Jump, 25m Sprint and Muscle Strength of hamstrings and Quadriceps), and a short warm-up program, followed by repeating the same tests as executed in baseline. The experimental group will receive Blood Flow Restriction within the warm-up routine, whereas the control group will do the same warm up program but without BFR.

On a separate occasion, the same athletes will perform the same warm-up routine with a Shear Wave Elastographic assessment of the Biceps Femoris Long Head before and after (immediately after, after 5 minutes and once more after 10 minutes) the warm-up.

ELIGIBILITY:
Inclusion Criteria:

* Free of pain at the moment of testing
* Adult (18+)
* Athletes (competitive team sport)

Exclusion Criteria:

* History of a hamstring strain injury
* History of cardiovascular problems
* Recent (<1 year) trauma or surgery of the lower extremity
* Reduced functioning or pain in the lower extremity.
* Not being able to perform physical activities, for whatever (medical) reason.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Change in muscle stiffness | (1) Before the warm-up routine, (2) immediately after the warm-up routine, (3) 5 minutes after the warm-up routine, and (4) 10 minutes after the warm-up routine
  The stiffness of the Biceps Femoris Long Head of the dominant leg will be assessed via a Shear Wave Elastography Device (Mach 30, SuperSonic Imagine), before and immediately after the warm-up routine. The muscle stiffness will be expressed in Kilopascals (kPa).
Change in jump height | (1) Before the warm-up routine and (2) immediately after the warm-up routine
  The jump height will be assessed during 5 consecutive countermovement jumps. This will be assessed with an OptoJump device. The highest jump will be taken into account. The jump height will be expressed in cm.
Change in muscle strength | (1) Before the warm-up routine and (2) immediately after the warm-up routine
  Muscle strength of the Hamstrings and Quadriceps muscles. Measured via a Hand Held Dynamometer. Strength will be expressed in Newton (N).
Change in sprinting speed | (1) Before the warm-up routine and (2) immediately after the warm-up routine
  Sprinting speed will be assessed at 5m, 10m and 25m. This via the use of timing gates. This outcome measure will be expressed in seconds (s).

SECONDARY OUTCOMES:
level of readiness | Immediately after the warm-up
  Participants will be asked after the warm-up (with or without BFR) how well they feel prepared to substitute into the game on a scale from 0-100; being zero = not ready at all, 100 = totally ready
Change in heart rate | (1) Right before the warm up, (2) after one minute, (3) after two minutes, (4) after 3 minutes, (5) at the end of the warm up
  This parameter will be captured to track the cardiovascular answer of the body during the warm-up by using a polar watch and elastic strap with a monitor around the waist.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Witvrouw, Principal Investigator — Departement of Rehabilitation Sciences, Ghent University
Locations (1):
- Ghent University, Ghent, Belgium